CLINICAL TRIAL: NCT05962229
Title: Comparative Pharmacokinetics and Pharmacodynamics of Synthetic Nicotine
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 22-36348; 1R01DA057282-01 (NIH)
Record Dates: First submitted 2023-07-17; First posted 2023-07-27 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Nicotine Dependence; Nicotine Vaping
Keywords: Nicotine Pharmacokinetics; Nicotine Pharmacodynamics; Vaping; E-cigarettes
MeSH Terms: conditions — Tobacco Use Disorder; Vaping | interventions — Nicotine; nicotine 1-N-oxide

STUDY DESIGN:
Intervention Model Description: Within-subject, single-blinded crossover study. Participants will be randomized to the order of the 3 conditions using a Latin Square design.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- S-nicotine (tobacco) as the starting condition (Experimental): Participants will spend 8 hours in the hospital research ward where they will vape e-liquid containing 100% (S)-nicotine.
  Interventions: Drug: (S)-Nicotine; Drug: (R)- nicotine; Drug: Racemic nicotine
- R-nicotine (synthetic) as the starting condition (Experimental): Participants will spend 8 hours in the hospital research ward where they will vape e-liquid containing 100% (R)-nicotine.
  Interventions: Drug: (S)-Nicotine; Drug: (R)- nicotine; Drug: Racemic nicotine
- Racemic (50:50 S- and R- nicotine) as the starting condition (Experimental): Participants will spend 8 hours in the hospital research ward where they will vape e-liquid containing 50% (S)-nicotine and 50% (R)-nicotine.
  Interventions: Drug: (S)-Nicotine; Drug: (R)- nicotine; Drug: Racemic nicotine

INTERVENTIONS:
Drug: (S)-Nicotine — Participants will spend 8 hours in the hospital research ward and will vape e-liquid containing 100% (S)-nicotine. They will vape following a standardized session, followed by a 4 hour abstinence period. Participants will then vape as they wish (ad libitum) for 90 minutes.
Drug: (R)- nicotine — Participants will spend 8 hours in the hospital research ward and will vape e-liquid containing 100% (R)-nicotine. They will vape following a standardized session, followed by a 4 hour abstinence period. Participants will then vape as they wish (ad libitum) for 90 minutes.
Drug: Racemic nicotine — Participants will spend 8 hours in the hospital research ward and will vape e-liquid containing 50% (R)-nicotine and 50% (S)-nicotine. They will vape following a standardized session, followed by a 4 hour abstinence period. Participants will then vape as they wish (ad libitum) for 90 minutes.
  Other Names: 50:50 mixture of (S)- and (R)-nicotine

SUMMARY:
In a crossover study, experienced electronic cigarette users will vape 3 different forms of nicotine: natural (derived from tobacco), synthetic, or a 50:50 mixture of both natural and synthetic. The investigators will compare nicotine metabolism, cardiovascular effects, patterns of self-administration, and participants' feelings of craving/withdrawal and enjoyment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy on the basis of medical history and limited physical examination.
* Current regular user of E-Cigarettes (≥ 15 days in the past 30 days)

Exclusion Criteria:

* • Medications

  * Use of medications that are inducers of nicotine metabolizing enzyme CYP2A6 (Example: rifampicin, carbamazepine, phenobarbital, and other anticonvulsant drugs).
  * Use of sympatholytic medications for cardiovascular conditions including hypertension (Example: beta and alpha-blockers).
  * Concurrent use of nicotine-containing medications (Example: nicotine patch, lozenge, gum).
  * Any stimulant medications (example: Adderall) generally given for ADHD treatment.

    • Pregnancy
  * Pregnancy (self-reported and urine pregnancy test)
  * Breastfeeding (determined by self-report)
  * Women of childbearing potential must be using an acceptable method of contraception

    * Inability to read and write in English
    * A known propylene glycol/vegetable glycerin allergy
    * Uncomfortable with getting blood drawn

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-12-06 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Mean Nicotine Exposure Over Time | Up to 7 hours
  Plasma nicotine area under the concentrated time curve (AUC) (ng/ml*h)

SECONDARY OUTCOMES:
Mean Amount of Nicotine Consumed Over Time | 120 minutes
  Nicotine self-administration determined by device weight change before and after use multiplied by the nicotine concentration in the e-liquid

CONTACTS AND LOCATIONS:
Overall Officials: Neal Benowitz, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Zuckerberg San Francisco General Hospital (ZSFG), San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No